CLINICAL TRIAL: NCT01748396
Title: Effect of Phosphate Binders on FGF-23 During Calcitriol Administration in CKD Stage 3 Patients
Brief Title: Effect of Phosphate Binders on FGF-23 With Concurrent Calcitriol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yon Su Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUH-FGF23
Record Dates: First submitted 2012-12-08; First posted 2012-12-12 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Kidney Disease Stage 3
Keywords: FGF-23; Calcitriol; Calcium carbonate; CKD Stage 3
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Calcitriol; Calcium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calcitriol + CaCO3 (Experimental): Calcitriol 0.25mcg 1cap daily for 8 weeks, and Calcium Carbonate 500mg 1tab 3 times daily for 8 weeks
  Interventions: Drug: Calcitriol; Drug: Calcium Carbonate
- Calcitriol (Active Comparator): Calcitriol 0.25mcg 1cap daily for 8 weeks
  Interventions: Drug: Calcitriol

INTERVENTIONS:
Drug: Calcitriol
Drug: Calcium Carbonate
  Arms: Calcitriol + CaCO3

SUMMARY:
Chronic kidney disease (CKD) is an established risk factor for cardiovascular morbidity and mortality, as shown by common manifestations of left ventricular hypertrophy (LVH) and arterial calcifications in CKD patients. Fibroblast growth factor-23(FGF-23) is a recently identified phosphaturic hormone that has been reported to be associated with the development of secondary hyperparathyroidism, cardiovascular morbidity, mortality, CKD progression.

While vitamin D is the mainstay therapy in CKD mineral bone disease (CKD-MBD), increased FGF-23 levels have been reported with vitamin D administration. The purpose of this study was to investigate the effect of calcium carbonate when used in conjunction with calcitriol on FGF-23.

ELIGIBILITY:
Inclusion Criteria:

* Adults of 18~70 years of age
* CKD stage 3 patients (GFR: 30-60ml/min/1.73m2)
* Patients who've given consent to the trial

Exclusion Criteria:

* Known allergy to Vitamin D or calcium carbonate
* Administration of vitamin D analogue or phosphate binders 3 months prior to study entry
* History of hypercalcemia (corrected serum calcium > 10.5 mg/dL) or hypophosphatemia (serum phosphate < 2.5 mg/dL) 3 months prior to study entry
* Patients with bone pathologies or diseases requiring vitamin D therapy that is unrelated to CKD-MBD
* Administration of concurrent medication , diseases, or history of surgeries that may affect bone-mineral metabolism or alter bone status
* Patients diagnosed with rapidly progressive glomerulonephritis(RPGN) or those in need of renal replacement therapy
* Patients with obstructive bowel diseases, or severe gastrointestinal diseases
* Patients with less than 2 years of life expectancy(ex. Malignancy diseases)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Percent changes in FGF-23 | 8 weeks after administration
  Comparison of percent changes in FGF-23 from baseline

SECONDARY OUTCOMES:
Percent changes in Ca | 8 weeks after administration
  Comparison of percent change in Ca from baseline
Percent changes in P | 8 weeks after administration
  Comparison of percent change in P from baseline
Percent changes in iPTH | 8 weeks after administration
  Comparison of percent change in intact parathyroid hormone from baseline
Percent changes in 25(OH)D | 8 weeks after administration
  Comparison of percent change in 25(OH)D from baseline
Percent changes in 1,25(OH)2D | 8 weeks after administration
  Comparison of percent change in 1,25(OH)2D from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Yon Su Kim, M.D., Ph.D., Principal Investigator — Seoul National University Hospital; Jung Mi Oh, Pharm.D., Study Chair — College of Pharmacy, Seoul National University
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086